CLINICAL TRIAL: NCT04524078
Title: Integrated Care Improves Risk-factor Modification After Transient Ischemic Attack or Minor Stroke Patients (Lleida TIA Intervention Study)
Brief Title: Lleida TIA Intervention Study
Acronym: LLETIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Francisco Purroy, Principal investigator, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LLETIS 1.0
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Transient Ischemic Attack
Keywords: transient ischemic attack
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: intensive integrated intervention care program [ICP] (lifestyle changes, patient education, adherence to practical guidelines) to transient ischemic attack or minor stroke patients would modify a variety of vascular risk factors and therefore should decrease the likelihood of recurrent stroke or vascular events
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive integrated intervention care program (Experimental): intensive integrated intervention care program [ICP] (lifestyle changes, patient education, adherence to practical guidelines) to transient ischemic attack or minor stroke patients would modify a variety of vascular risk factors and therefore should decrease the likelihood of recurrent stroke or vascular events
  Interventions: Other: intensive integrated intervention care program
- Non intensive integrated intervention care program (No Intervention)

INTERVENTIONS:
Other: intensive integrated intervention care program — intensive integrated intervention care program [ICP] (lifestyle changes, patient education, adherence to practical guidelines) to transient ischemic attack or minor stroke patients would modify a variety of vascular risk factors and therefore should decrease the likelihood of recurrent stroke or vascular events
  Arms: Intensive integrated intervention care program

SUMMARY:
Having a transient ischemic attack (TIA) or a minor stroke is a real risk factor not only for early recurrent stroke but also for major extracranial vascular events. Despite these warning events provide an opportunity for prevention usual post-discharge care of these subjects (mainly at primary care) is not associated with an optimal control of cerebrovascular risk factors (CRF). The investigators hypothesized that patients exposed to the intensified integrated multifactorial interventional care program (ICP) model would exhibit better management of CRF and receive more targeted advice than patients receiving standard care. A second objective was to investigate the effect of the ICP model on stroke recurrence or the appearance of major extracranial vascular events.

To test this hypothesis the investigators perform a controlled, randomized, single blind, parallel trial. Subjects are recruited at the Stroke Unit and are randomized into two groups: 1. usual care (control group) and 2. ICP (intervention group). Patients assigned to receive usual care (general practitioner with the possibility of being referred to specialists) are compared to those assigned to undergo ICP. This ICP involves strict treatment goals (LDL-cholesterol <100 mg/dl, blood pressure <130/80 mmHg, HbA1c<7%, no smoking, regular exercise and no excessive alcohol consumption) to be achieved through behavior modification (diet, physical activity, smoking cessation, alcohol cessation) and a stepwise introduction of pharmacologic therapy for the main CRF (hypercholesterolemia, hypertension and diabetes). This multifactorial intervention is overseen in each primary care center by a trained general practitioner and nursery. The treatment goals are the same for the control group and the intervention group. General practitioners caring patients of each group are informed of these strict treatment goals. Patients in the ICP group receive a minimum of four scheduled individual consultations in one year (baseline, 3, 6 and 9 months). Primary and secondary outcomes are evaluated by an external Neurologist at 12 months after their inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with transient ischemic attack (reversible episode of neurological deficit of ischemic origin that resolved completely within 24 hours) or minor stroke (established neurological deficit of ischemic origin with US National Institutes of Health stroke scale [NIHSS]score of 3 or less at the time of randomization)
2. All subjects will be clinically evaluated by a stroke neurologist
3. All subjects will be evaluated with CT scan or MRI to exclude other causes of neurological symptoms different than brain ischemia
4. Patients with independence: modified Rankin score<3
5. Patients with a critical carotid stenosis will be included after revascularization therapy
6. Written informed consent

Exclusion Criteria:

1. Having serious comorbidities: dementia, advanced Cancer, excessive intake of alcohol (> 280 gr/week), severe renal or hepatic insufficiency and severe cardiac failure
2. Currently receiving an investigational drug or device
3. Age<18 years
4. Patient or family declining to take part
5. Pregnant or breastfeeding
6. Transient neurological deficit for < 5 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Controlled blood pressure | 12 months
  Rate of patients with controlled blood pressure values (Systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg) and controlled LDL-c (levels <100 mg/dl)
Controlled LDL levels | 12 months
  Rate of patients with controlled LDL-c (levels <100 mg/dl)

SECONDARY OUTCOMES:
Stroke recurrence | 12 months
  Rate of patients with stroke recurrence
Stroke recurrence | 5 years
  Rate of patients with stroke recurrence
Stroke recurrence | 10 years
  Rate of patients with stroke recurrence
Major vascular events | 12 months
  Rate of patients with stroke recurrence
Major vascular events | 5 years
  Rate of patients with stroke recurrence
Major vascular events | 10 years
  Rate of patients with stroke recurrence